CLINICAL TRIAL: NCT03588845
Title: Pragmatic, Multicenter, Cluster, Cohort Randomized Controlled Treat-to-target Trial for Treatment of SIBO in SSc Pilot
Brief Title: The Small Intestine Bacterial Overgrowth Study Pilot
Acronym: SIBO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canadian Scleroderma Research Group (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Murray Baron, Dr., Canadian Scleroderma Research Group
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CODIM-MBM-16-282
Record Dates: First submitted 2018-05-10; First posted 2018-07-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Systemic Sclerosis; Small Intestinal Bacterial Overgrowth
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Clinical Protocols; Standard of Care

STUDY DESIGN:
Intervention Model Description: The primary objective of this randomized trial is to determine if a structured, treat-to-target algorithm based on treatment response and relapse performs better than standard care for the treatment of symptoms SSc-SIBO.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol Treatment (Other): If a score on the GSS is > 5, the computer will send an automatic notice to the office of the doctor and to the doctor him/herself telling them of this.
  Upon receipt of the notice, the protocol doctors will be expected to make an appointment within the timeframe outline in the protocol. Upon receipt of this notice the secretaries or clerks at the site will be asked to insert a treatment sheet in the doctor's chart. This sheet will be used to assess the timeliness of the first visit after notification, about the adherence of protocol doctors to protocol treatment.
  Interventions: Other: Treatment Protocol
- Standard of Care (Other): Standard care doctors, who will not know the details of this protocol, will decide on their own if and when to see the patient. Upon receipt of this notice the secretaries or clerks at the site will be asked to insert a treatment sheet in the doctor's chart. This sheet will be used to assess types of medications and general pattern of treatment of the standard of care doctors.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Treatment Protocol — Protocol treatment sites will be expected to see the patient within a pre-specified window of time. The doctors at that site will apply the treatment algorithm and will make decisions about response to treatment based on the algorithm and on specific patient answers to questionnaires. The treatment protocol will only be made available to IRBs, not to any site personnel before randomization. This was derived from a survey of rheumatologists in many countries and gastroenterologists, mostly in North America, who were asked multiple questions about how they would treat and follow up patients with suspected SIBO. Successful treatment is a response on GSS of no diarrhea plus a total GSS of < 5.
  Arms: Protocol Treatment
Other: Standard of Care — Physicians randomly assigned to standard of care will also be informed of their patients who met eligibility criteria. They will not be aware of the detailed treatment protocol but will be informed of which medications are in the protocol eg antibiotics, prokinetics etc. They will be free to contact the patients at their convenience and to treat them in any way they deem suitable, preferably using these medications but at doses and frequencies according to their own wishes.
  Arms: Standard of Care

SUMMARY:
This is a pragmatic study in which will compare a detailed treat-to-target (T2T) treatment algorithm to standard care for SSc SIBO at multiple sites around the world. The treatment algorithm was developed from the results of a survey of SIBO treatment preferences of rheumatologists and gastroenterologists. Although the drugs in the algorithm are already used in SSc, there is no uniform way of doing this and assessing the patient response. A very standardized protocol was created with details of how to use the medications, the duration of use and the timing of different drugs. In addition, symptoms of SIBO will be dectected by having patients complete a validated screening questionnaire, the global symptomatic score (GSS), online every 3 months for the duration of the study. A score > 5 is very strongly related to bacterial overgrowth. In other studies, about 40% of unselected patients score at this level. This same questionnaire will be used in the T2T doctors' offices to decide if response is adequate and will also be used to assess outcome in the algorithm group versus standard care group.

The primary outcome is the change in symptoms based on the total GSS. Secondary outcomes will include examination of all GSS subscales. HRQoL will be assessed by the social scale of the newly developed UCLA SSc GIT 2.0 questionnaire, which has become the standard GI questionnaire in SSc trials.

￼￼￼RN. # 00296313

DETAILED DESCRIPTION:
Objectives: To determine the feasibility of the full project. This will be a trial with 3 months of recruitment and 6 months of follow up for each case.

Specific Aims:

1. Determine if REBs perceive any major issues regarding the full trial.
2. Determine if the sites are consenting all eligible patients.
3. Determine the signing rate of consent.
4. Determine patient adherence to web access for questionnaires.
5. Assess the method for detecting eligible cases from web questionnaires.
6. Assess whether physician notifications are being sent out quickly after detecting eligible cases.
7. Assess the timeliness and completeness of physician receipt of notification of patient eligibility.
8. Assess physician adherence to treatment protocol:

   1. how soon protocol patients are brought in to see doctor after receipt of notice.
   2. does doctor record what he does accurately.
   3. does he/she schedule return visits according to protocol.
   4. does he/she use in office questionnaires for treat to target.
   5. does he/she base decisions on these questionnaires.
   6. does he/she follow algorithm sequentially.
9. For control sites,

   1. Record how soon protocol patients are brought in to see doctor after receipt of notice.
   2. Assess whether the doctor accurately records what he/she does.

      10 international sites will be chosen from the INSYNC cohort located in Australia, Canada, the U.S., the Netherlands, Spain, Germany and Sweden. In each country one site will be randomly selected to be a protocol site and one standard care site. This selection will provide representation from English and non-English speaking centres and from an array of countries with different medical cultures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Scleroderma
* Internet access
* An email address
* Adequate computer literacy in order to fill out the online questionnaires.

Exclusion Criteria:

* Allergy to protocol drugs
* Concomitant disease that would make it unlikely that they will survive for one year
* Use of substances known to cause diarrhea
* History of antibiotics in the 12 weeks prior to inclusion
* History of intestinal pseudo-obstruction
* Inability to complete the symptom questionnaires
* No functional level of written & spoken languages
* Previous C. Dificile infection
* Previous gastrointestinal surgery
* Prolonged QT interval
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Determine if protocol treatment is effective | 3 years
  The primary outcome is the total Gastrointestinal Symptom Scale score. Each symptom carries a score from 0 (no symptoms) to 3 (severe). The maximum overall score is 33. An improvement in the score, ie a lower score, indicates an improvement in GI symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- John's Hopkins, Baltimore, Maryland, United States
- Saint Vincent's, Melbourne, Australia

DOCUMENTS (1):
  • Study Protocol (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT03588845/Prot_000.pdf